CLINICAL TRIAL: NCT00555308
Title: Emergency Department Targeted Ultrasound for the Detection of Hydronephrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Dr. Kieran Moore, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EMED 094-07; PSI Grant Sept 2007
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Urolithiasis; Ultrasonography; Hydronephrosis
Keywords: urolithiasis; ultrasound; hydronephrosis
MeSH Terms: conditions — Urolithiasis; Hydronephrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one (Experimental): undergo EDTU
  Interventions: Other: emergency department targeted ultrasound imaging

INTERVENTIONS:
Other: emergency department targeted ultrasound imaging — bedside ultrasound performed by emergency physician to identify hydronephrosis
  Other Names: EDTU

SUMMARY:
An Emergency Department Targeted Ultrasound (EDTU) is an ultrasound examination performed by an emergency department physician, instead of a radiologist or ultrasound technician. EDTU is intended to be a readily assessable test performed at the bedside, to quickly and safely determine the presence of a disease state; it answers a binary question, as compared to formal ultrasound imaging which seeks to determine the cause of a patient's symptoms.

The objective of this study is to determine the accuracy of EDTU in patients suspected of renal colic. By demonstrating excellent test characteristics, these investigators hope that this research will be used to incorporate EDTU for hydronephrosis into standard emergency care in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department patients
* Males and Females
* Age 16-65
* Undergoing CT scan of the abdomen or formal ultrasound of the abdomen at Kingston General Hospital or Hotel Dieu Hospital in Kingston, Ontario.

Exclusion Criteria:

* Hemodynamic instability
* Fever
* Leukocytes or nitrites on dipstick urinalysis
* Pregnancy
* Renal failure
* Single functioning kidney or renal transplant

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of EDTU | 1 hour

SECONDARY OUTCOMES:
same measures of diagnostic accuracy in the planned subgroup of patients being investigated for suspected renal colic | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Bruder, MD, Principal Investigator — Queen's University; Kieran M Moore, MD MMSc, Study Director — Queen's University; Louise Rang, MD RDMS, Study Director — Queen's University
Locations (2):
- Canada (2):
  - Hotel Dieu Hospital, Kingston, Ontario
  - Kingston General Hospital, Kingston, Ontario